CLINICAL TRIAL: NCT05717166
Title: A Randomized Phase III Trial of Stereotactic Ablative Radiotherapy for Patients With Up to 10 Oligometastases and a Synchronous Primary Tumor.
Acronym: SABR-SYNC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: David Palma (Other)
Responsible Party: Sponsor-Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ReDA 13176
Record Dates: First submitted 2023-01-26; First posted 2023-02-08 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Drug Therapy; Immunotherapy; Observation; Surgical Procedures, Operative; Radiofrequency Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm (Arm 1) (Active Comparator): Radiotherapy for patients in the standard arm should follow the principles of palliative radiotherapy as per the individual institution, with the goal of alleviating symptoms or preventing imminent complications.
  Interventions: Radiation: Palliative Radiotherapy; Drug: Chemotherapy; Drug: Hormone therapy; Drug: Immunotherapy; Drug: Targeted Systemic Therapy; Other: Observation
- Experimental Arm (Arm 2) (Experimental): Consists of treatment to the primary tumor and metastases, with SABR preferred, but other options all allowable (e.g. surgery, RFA, fractionated radiation, chemoradiation) if those are deemed to be preferable by the treating oncologists.
  Interventions: Radiation: Palliative Radiotherapy; Drug: Chemotherapy; Drug: Hormone therapy; Drug: Immunotherapy; Drug: Targeted Systemic Therapy; Other: Observation; Radiation: Stereotactic Ablative Radiotherapy; Procedure: Surgery; Other: Radiofrequency Therapy (RFA); Radiation: Fractionated Radiation

INTERVENTIONS:
Radiation: Palliative Radiotherapy — Radiotherapy for patients in the standard arm should follow the principles of palliative radiotherapy as per the individual institution, with the goal of alleviating symptoms or preventing imminent complications. Recommended dose fractionations in this arm will include 8 Gy in 1 fraction, 20 Gy in 5 fractions, and 30 Gy in 10 fractions.
Drug: Chemotherapy — Pre-specified based on the standard of care approach for that patient.
  Other Names: Cytotoxic Systemic Therapy
Drug: Hormone therapy — Pre-specified based on the standard of care approach for that patient.
  Other Names: Hormonal Systemic Therapy
Drug: Immunotherapy — Pre-specified based on the standard of care approach for that patient.
Drug: Targeted Systemic Therapy — Pre-specified based on the standard of care approach for that patient.
Other: Observation — Pre-specified based on the standard of care approach for that patient.
Radiation: Stereotactic Ablative Radiotherapy — The primary tumor may be treated with SABR or with other local modalities at the discretion of the treating team and/or the local multidisciplinary tumor board.
  Preferred doses are 20 Gy in 1 fraction, 30 Gy in 3 fractions (every second day), and 35 Gy in 5 fractions (daily).
  Arms: Experimental Arm (Arm 2)
Procedure: Surgery — Treatment to the primary tumor and metastases, with SABR preferred, but other options all allowable if those are deemed to be preferable by the treating oncologists.
  The primary tumor may be treated with SABR or with other local modalities at the discretion of the treating team and/or the local multidisciplinary tumor board. Because of the convenience in using SABR for all lesions, non-SABR modalities should only be used if they are likely to provide a benefit over SABR.
  Arms: Experimental Arm (Arm 2)
Other: Radiofrequency Therapy (RFA) — Treatment to the primary tumor and metastases, with SABR preferred, but other options all allowable if those are deemed to be preferable by the treating oncologists.
  Arms: Experimental Arm (Arm 2)
Radiation: Fractionated Radiation — Treatment to the primary tumor and metastases, with SABR preferred, but other options all allowable if those are deemed to be preferable by the treating oncologists.
  Tumors in the esophagus, stomach, small intestine or colon should be treated with either fractionated radiation or a lower SABR dose (e.g. 25 Gy in 5 fractions) to minimize the risk of perforation.
  Arms: Experimental Arm (Arm 2)

SUMMARY:
This study is a phase III multi-institutional randomized trial. Patients will be randomized in a 1:2 ratio between current standard of care treatment (Arm 1) vs. standard of care treatment + SABR (Arm 2) to sites of known disease.

Patients will be stratified by two of the strongest prognostic factors, based on a large multi-institutional analysis3: histology (Group 1: hormone-sensitive prostate cancer, breast, or renal; Group 2: all others), and number of metastases (Group 1: 1-3; Group 2: 4-10).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Willing to provide informed consent
* Karnofsky performance status > 60
* Life expectancy > 6 months
* Histologically confirmed malignancy with metastatic disease detected on imaging. Biopsy of metastasis is preferred, but not required.
* Total number of metastases 1-10 at the time of enrollment, with a primary tumor also present
* Restaging completed within 12 weeks prior to randomization (see section 5.1)
* For patients receiving thoracic radiotherapy, the enrolling physician must confirm there are no computed tomography (CT) changes suggestive of fibrotic interstitial lung disease (ILD) (i.e. reticular changes, traction bronchiectasis, or honeycombing) reported on any prior CT scans. If any are present, the patient must be assessed by a respirologist to rule out ILD prior to enrollment.
* 10 or fewer lifetime metastases from the cancer for which participants are being enrolled

Exclusion Criteria:

* Serious medical comorbidities precluding radiotherapy. These include ILD in patients requiring thoracic radiation, Crohn's disease in patients where the gastrointestinal (GI) tract will receive radiotherapy, or ulcerative colitis where the bowel will receive radiotherapy and connective tissue disorders such as lupus or scleroderma.
* For patients with liver metastases, moderate/severe liver dysfunction (Child Pugh B or C); please see the Child-Pugh score calculator.
* Substantial overlap with a previously treated radiation volume. Prior radiotherapy in general is allowed, as long as the composite plan meets dose constraints herein. For patients treated with radiation previously, biological effective dose calculations should be used to equate previous doses to the tolerance doses listed in Appendix 1. All such cases must be discussed with a member of the study steering committee.
* Malignant pleural effusion
* Inability to treat all sites of disease
* Brain metastasis > 3 cm in size or a total volume of brain metastases greater than 30 cc.
* Metastasis in the brainstem
* Clinical or radiologic evidence of spinal cord compression
* Metastatic disease that invades any of the following: GI tract (including esophagus, stomach, small or large bowel), or skin
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Approximately end of year 6 (Study Completion)
  Time from randomization to death from any cause, or date of last follow-up, whichever occurs first.

SECONDARY OUTCOMES:
Quality of Life (QOL) assessed with the Functional Assessment of Cancer Therapy: General (FACT-G). | Quality of Life outcomes to be collected for the first 2 years (3, 6, 12, 18, 24 months)
Quality of Life (QOL) assessed with the Functional Assessment of Cancer Therapy: The EuroQol 5-Dimension 5-Level (EQ-5D-5L). | Quality of Life outcomes to be collected for the first 2 years (3, 6, 12, 18, 24 months)
Toxicity assessed by the Common Toxicity Criteria for Adverse Events (CTCAE) version 5 for each organ treated (e.g. liver, lung, bone). | Toxicity outcomes to be collected for the first 2 years (Last week of treatment, in 6 weeks, in 3, 6, 12, 18, 24 months)
Time to next systemic therapy | From randomization to year 6 (study completion).
  The time from randomization until commencement of any systemic anti-cancer therapy, or date of last follow-up, whichever occurs first.
Receipt of additional radiation during follow-up | During year 6 (follow-up year).
  Will be collected for SABR (as a binary endpoint; yes/no), and non-SABR (yes/no).

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (4):
  - BC Cancer - Centre for the North, Prince George, British Columbia
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario
  - Centre Hospitalier de l'Université de Montréal-CHUM, Montreal, Quebec
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palma DA, Giuliani ME, Correa RJM, Schneiders FL, Harrow S, Guckenberger M, Zhang T, Bahig H, Senthi S, Chung P, Olson R, Lock M, Raman S, Bauman GS, Lok BH, Laba JM, Glicksman RM, Nguyen TK, Lang P, Helou J, Goodman CD, Mendez LC, van Rossum PSN, Warner A, Gaede S, Allan AL. A randomized phase III trial of stereotactic ablative radiotherapy for patients with up to 10 oligometastases and a synchronous primary tumor (SABR-SYNC): study protocol. BMC Palliat Care. 2024 Sep 7;23(1):223. doi: 10.1186/s12904-024-01548-7. PMID 39244532